CLINICAL TRIAL: NCT02662062
Title: Pembrolizumab With Chemoradiotherapy as Treatment for Muscle Invasive Bladder Cancer
Acronym: PCR-MIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 1502
Record Dates: First submitted 2016-01-13; First posted 2016-01-25 (Estimated); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-05

CONDITIONS: Bladder Cancer
Keywords: Non-metastatic muscle invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab to be administered via IV 200mg 3 weekly commenced concurrently with chemoradiotherapy, and continuing until 12 week cystoscopy.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg/m2, IV (in the vein) on day 1 every three weeks (Weeks 1, 3, 7, 10, 13, 16 and 19). until progression or unacceptable toxicity develops.
Drug: Cisplatin — 35 mg/m2, IV (in the vein) every week for six weeks.
Radiation: Radiotherapy — 2.00Gy once daily for 32 fractions, 5 fractions/week over six weeks and two days (a total of 64Gy).

SUMMARY:
This study will enrol patients with maximally resected (via transurethral resection (TURBT) non-metastatic muscle invasive bladder cancer, who either wish to attempt bladder preservation therapy or are ineligible for cystectomy. Patients must have adequate organ function and performance status to receive cisplatin based chemoradiotherapy, and no contraindications to the use of pembrolizumab. The study will enrol 30 patients to be treated with pembrolizumab and radiotherapy.

All patients will be planned to be treated with 64Gy of radiation therapy in 32 fractions over 6 weeks and 2 days. All patients will receive cisplatin 35mg/m2 IV concurrently weekly with radiation therapy for 6 doses total. Pembrolizumab will commence concurrently with radiation and be given 200mg IV every 21 days, continuing until the 12 week cystoscopy and assessment.

Surveillance cystoscopy will be performed 12 weeks after the commencement of chemoradiotherapy, and assess the rate of complete response to therapy. A safety follow up visit will occur 4 and 12 weeks post cystoscopy. From week 31 survival follow up will commence with clinical assessment, cystoscopy and CT staging performed at intervals until 5 years.

The objective of the study is to assess the safety and feasibility of combining pembrolizumab with chemoradiotherapy. The primary endpoint assessed will be safety, as defined by a satisfactorily low rate of unacceptable toxicity (G3-4 adverse events or failure of completion of planned chemotherapy and radiotherapy according to defined parameters). The secondary endpoint will be efficacy, as assessed by complete response rate of the primary tumour at first post chemoradiotherapy cystoscopic assessment. Exploratory analysis will include assessment of tumour histopathological, molecular, genetic and immunological parameters.

It is expected that it will take two years to accrue the required 30 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have histologically-confirmed diagnosis of muscle-invasive T2-T4a, Nx or N0 urothelial cell carcinoma of the bladder. Subjects with tumors of mixed transitional/non-transitional cell histology are allowed, but transitional cell carcinoma must be the predominant histology (>50%). Subjects with predominant or exclusively non-transitional cell histology are not allowed.
4. Must have undergone maximal transurethral resection of the bladder tumour, as is judged as safe as possible by the urologist performing the resection, within 42 days of treatment. Where patient has only had a biopsy/partial resection and is otherwise eligible for entry into the study, the case should be rediscussed with the referring urologist to see whether further resection would be feasible prior to embarking with the chemo-radiotherapy.
5. Have elected not to undergo radical cystectomy, or are unsuitable for radical cystectomy.
6. Planned for chemoradiotherapy as definitive treatment.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale
8. Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days of registering the patient on the trial.

   * Absolute neutrophil count (ANC): ≥1.5 X 10^9/L
   * Platelets: ≥100 X 10^9/L
   * Hemoglobin: ≥9 g/dL without transfusion or EPO dependency
   * Calculated creatinine clearance ≥50 mL/min
   * Serum total bilirubin: ≤ 1.5 X ULN OR
   * Direct bilirubin ≤ ULN for participants with total bilirubin levels: > 1.5 ULN
   * AST and ALT: ≤ 2.5 X ULN
   * Albumin: >25 g/dL
   * International Normalized Ration (INR) or Prothrombin Time (PT): ≤1.5 X ULN unless participant is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
   * Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN unless participant is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
9. Female participant of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registering the patient. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female participants of childbearing potential should be willing to use two methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
12. Willing to consent to the use of their collected tumour specimen, blood and urine as detailed in the protocol for future scientific research including but not limited to DNA, RNA and protein based biomarker detection.

Exclusion Criteria:

1. Has concurrent extra-vesical (i.e. urethra, ureter or renal pelvis) urothelial cell carcinoma of the urothelium. Patients who have involvement of the prostatic urethra with urothelial cell cancer (TCC) that was visibly completely resected and no evidence of stromal invasion of the prostate remain eligible.
2. Evidence of tumour-related moderate/severe hydronephrosis unless stented or with nephrostomy to preserve renal function.
3. Extensive or multifocal bladder carcinoma in situ (CIS) precluding curative chemoradiotherapy.
4. Bulky T3/T4a tumours unsuitable for curative treatment (i.e. >10 cms in any dimension); node positive disease
5. Evidence of distant metastatic disease on CT chest/abdomen/pelvis performed within 42 days prior to study entry. Patients with pelvic lymph nodes deemed to be 'positive' are not eligible for the study unless histological confirmation of the largest most suspicious node is negative for malignancy. Patients with known CNS metastatic disease are excluded from the study
6. Prior pelvic radiotherapy
7. Has had prior intravenous chemotherapy, targeted small molecule therapy, or radiation therapy for treatment of bladder cancer. Prior intravesical use of BCG and mitomycin is permissible.
8. Unsuitable for concurrent cisplatin based chemoradiotherapy based on:

   * CTCAE v.4.03, Grade >2 audiometric hearing loss (25dB in two consecutive wave ranges) if previously performed.
   * CTCAE v.4.03, Grade >2 peripheral neuropathy
9. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of treatment.
10. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to registering the patient. Patients with adrenal insufficiency receiving replacement dose steroids are allowed on the trial.
11. Has a known history of active TB (Bacillus Tuberculosis)
12. Hypersensitivity to pembrolizumab or any of its excipients.
13. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
14. Prior or concurrent known additional malignancy of any site unless disease free for 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, Stage T1a well differentiated prostatic carcinoma in men (Gleason = 3+3, PSA <5)
15. Has any history of active autoimmune disease, Stevens-Johnson syndrome or Guillain-Barre. Exceptions to this are:

    * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone.
    * Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen who are also be eligible for this study.
16. Has known history of, or any evidence of active, non-infectious pneumonitis.
17. Has an active infection requiring systemic therapy.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
21. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
22. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
23. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
24. Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farshad Foroudi, MBBS, Principal Investigator — Austin Health; Nathan Lawrentschuk, MBBS, Principal Investigator — Austin Health
Locations (7):
- Australia (7):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weickhardt A, Foroudi F, Lawrentschuk N, Xie J, Sidhom M, Pal A, Grimison P, Zhang A, Ng S, Tang C, Hovey E, Chen C, Hruby G, Guminski A, McJannett M, Conduit C, Tran B, Davis ID, Hayne D. Pembrolizumab with Chemoradiation as Treatment for Muscle-invasive Bladder Cancer: Analysis of Safety and Efficacy of the PCR-MIB Phase 2 Clinical Trial (ANZUP 1502). Eur Urol Oncol. 2024 Jun;7(3):469-477. doi: 10.1016/j.euo.2023.09.011. Epub 2023 Oct 7. PMID 37806844
- See also: Sponsor's website — http://www.anzup.org.au

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 28
Completed | 27
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 72 [58 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 28
ECOG [Count of Participants; unit: Participants] — ECOG performance status scale describes a patients level of functioning in terms of their ability to care for themselves, daily activity and physical ability.
  Only participants ECOG 0-1 are eligible for this study. ECOG 0 - Fully active, able to carry on all pre-disease performance without restriction ECOG 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG 0 | 18
    ECOG 1 | 10
Histology [Count of Participants; unit: Participants]
  Transitional cell/ Urothelial | 25
  Mixed Transitional/ nontransitional | 3
  Associated carcinoma in situ | 9
T stage [Count of Participants; unit: Participants] — The T stage from the TNM classification describes the depth of invasion through the bladder wall and involvement of nearby tissues. All participants in this study were T2 or T3 with description below.
  T2 - The cancer has grown into the muscle layer of the bladder wall, but it has not passed completely through the muscle to reach the layer of fatty tissue that surrounds the bladder.
  T3 - The cancer has grown through the muscle layer of the bladder and into the layer of fatty tissue that surrounds the bladder it has not spread to surrounding tissues
  Participants
    T2 | 26
    T3 | 2
Prior BCG (Bacillis Calmette-Guerin vaccine) treatment [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing an Unacceptable Level of Toxicity as Defined Below
Description: Unacceptable toxicity was predefined as fitting one of the following categories.
  * Grade 3 or worse adverse event per CTCAE V 5.0 (excluding urinary adverse events Grade 3 and Grade 4)
  * Cisplatin is withheld for 2 or more doses
  * Cisplatin is withheld or dose reduced such that <66% of the intended total cisplatin dose is delivered
  * Radiation therapy extended beyond 7 weeks
  * Any single pembrolizumab dose is delayed for >6 weeks
Time Frame: 12 weeks of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
Participants
  Unacceptable toxicity - total | 9
  Grade 3 or higher adverse event | 6
  Immune mediated toxicity meeting unacceptable toxicity definition. | 2
  Cisplatin dose omissions 2 or greater | 4
  Radiation duration >7 weeks | 2
  Pembrolizumab >6 weeks delay | 1
Statistical Analysis 1: Comparison: Pembrolizumab; The null hypothesis is that the addition of pembrolizumab to chemoradiation is not unsafe (percentage of the population experiencing unacceptable toxicity is not >50%); Test type: Other — This is a single arm study looking at a binary value with the hypothesis suggesting it falls within a certain range; A Clopper-Pearson method was used to determine the unacceptable toxicity rate and a 95% confidence interval for this binary outcome measure

2. Secondary Outcome: Complete Response Rate at Week 19 of the Trial (12 Weeks Post Completion of Chemoradiotherapy).
Description: Complete response defined at this time point by fulfillment of all of the following criteria:
  i) the bi-manual examination under anesthesia is negative (performed at the time of cystoscopy) ii) All biopsies are negative for any tumor at the site(s) of pre-treatment tumor(s) iii) There is an absence of metastatic disease on most recently performed imaging of chest/abdomen and pelvis
Time Frame: Week 19 (12 weeks post chemotherapy)
Population: Only 21 patients were evaluable at this timepoint
Measure: Number (95% Confidence Interval); unit: Percentage of evaluable population
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
Percentage of evaluable population | 90 [70 to 99]
Statistical Analysis 1: Comparison: Pembrolizumab; Test type: Other — Single arm study with no comparator arm and assessment of a binary variable. Clopper-Pearson method used to calculate the 95% confidence interval relating to this proportion; Single arm study with no comparator arm and assessment of a binary variable. Clopper-Pearson method used to calculate the 95% confidence interval relating to this proportion

3. Secondary Outcome: The Complete Response Rate Assessed at Week 31 of the Trial (24 Weeks Post Completion of Chemoradiotherapy).
Description: as for outcome 2
Time Frame: Week 31 of the trial (24 weeks post completion of chemoradiotherapy)
Population: two participants not evaluable for this endpoint due to withdrawal of consent (1) and death from an exacerbation of pre-existing airways disease (1)
Measure: Number (95% Confidence Interval); unit: Percentage of evaluable population
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
Percentage of evaluable population | 88 [70 to 98]
Statistical Analysis 1: Comparison: Pembrolizumab; Test type: Other — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Estimated Median Overall Survival
Description: Estimation after characterization with a Kaplan Meier curve
Time Frame: median follow up 39 months
Population: 2 participants not evaluable for this endpoint due to withdrawal of consent (1) and death from pre-existing airways disease (1)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
months | 39 [17 to NA] — missing upper level of 95% confidence interval on the survival estimate from Kaplan-Meier estimator due to small number of events
Statistical Analysis 1: Comparison: Pembrolizumab; Test type: Other — Non comparative trial with a single arm; Kaplan Meier Estimate = 39, 95% CI 2-sided [lower limit 17] (missing upper limit of 95% confidence interval on the survival estimate from Kaplan-Meier estimator due to small number events)

5. Secondary Outcome: Overall Survival at 12 Months Post Study Entry
Description: Overall survival timepoint estimated after characterization on a Kaplan Meier curve
Time Frame: 12 months post study entry
Population: Two participants not evaluable for this endpoint due to withdrawal of consent (1) and death from pre-existing airways disease (1)
Measure: Number (95% Confidence Interval); unit: Percentage of evaluable population
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
Percentage of evaluable population | 92 [72 to 98]
Statistical Analysis 1: Comparison: Pembrolizumab; Test type: Other — Kaplan Meier Estimate performed for a 12 month timepoint in a single arm non comparative study; Kaplan Meier Estimate = 92, 95% CI 2-sided [72 to 98]

6. Secondary Outcome: Distant Metastasis Free Survival (DMFS) at 12 Months
Description: End point was characterized using a Kaplan Meier curve and 12 month time point assessed.
Time Frame: At 12 months post study entry
Population: 1 patient was not evaluable for this time point due to withdrawal of consent
  1 patient was not evaluable for this time point due to death related to pre-existing chronic airways disease
Measure: Number (95% Confidence Interval); unit: Percentage of population
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
Percentage of population | 85 [64 to 94]
Statistical Analysis 1: Comparison: Pembrolizumab; Test type: Other — Kaplan Meier Estimate of single arm non comparative study; Kaplan Meier Estimate = 85, 95% CI 2-sided [64 to 94]

7. Secondary Outcome: Local Disease Free Survival (LRPFS) at 12 Months
Description: Local recurrence was defined as recurrence in the bladder or a nodal recurrence in the pelvis
Time Frame: 12 months post therapy commencement
Population: Two participants not evaluable for this outcome measure for reasons of withdrawal of consent (1) and death from pre-existing airways disease (1)
Measure: Number (95% Confidence Interval); unit: Percentage of evaluable population
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
Percentage of evaluable population | 88 [68 to 98]
Statistical Analysis 1: Comparison: Pembrolizumab; Test type: Other — Kaplan Meier estimate at a 12 month timepoint for a single arm non comparative study; Kaplan Meier Estimate = 88, 95% CI 2-sided [68 to 98]

8. Other Pre Specified Outcome: The Abundance and Composition of Tumour Infiltrating Lymphocytes, as Assessed by Immunohistochemical Analysis, of Patients Pre-treatment Tissue Samples.
Description: Resected tumour specimens will be available from the patients enrolled on the trial. These pre-treatment specimens will be comprehensively profiled for the abundance and composition of tumour infiltrating lymphocytes (CD4, CD8, CD3, CD20 and FoxP3 positive cells) by immunohistochemistry using the state-of-the-art Vectra Automated Imaging system which enables multiplexed immunohistochemical analysis.
Time Frame: Through study completion, an average of 7 years.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in Gene Expression in CD3+ Cells Pre and Post-treatment as Assessed by RNAseq Analysis to Assess for Gene Expression Changes Associated With Immune Activation.
Time Frame: Through study completion, an average of 7 years.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in the Immune Regulatory Molecules OX-40/LAG3/PD1/ICOS on T Cell Subsets as Assessed by Flow Cytometry.
Description: Blood samples collected prior to treatment, at the end of chemoradiotherapy, and after 24 weeks will be collected from the patients on the trial. PBMCs will be isolated using Ficoll, and changes in specific immune subpopulations (number/ratio) determined by multi-parameter FACS. Changes in the immune regulatory molecules OX-40/LAG3/PD1/ICOS on T cell subsets will be assessed by flow cytometry.
Time Frame: Through study completion, an average of 7 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the period of enrollment in the study (Planned out to 5 years post commencement) the median follow up at the conclusion of the trial was 39 months
Description: Adverse events were collected at each visit during treatment and follow up and they were recorded per CTCAE Version 5.0
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 8/28
Serious Adverse Events (participants affected / at risk) | 13/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=28)
Urinary tract infection (Infections and infestations) | 2
Haematuria (Renal and urinary disorders) | 2
Fever (General disorders) | 2
Renal and urinary discorders (other) (Renal and urinary disorders) | 1 — Renal tract obstruction
Musculoskeletal and Conncective tissue disorder (other) (Musculoskeletal and connective tissue disorders) | 1 — Immune mediated muscoloskeletal pain
Hypetension (Vascular disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Infusion related reaction (Product Issues) | 1
Metabolism and nutritional disorder (other) (Metabolism and nutrition disorders) | 1 — Reported as an instance of Serotonin syndrome with Fevers, rigors, tachycardia and spasticity
Delusions (Psychiatric disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1 — Rib fracture
infections and infestations (other) (Infections and infestations) | 1 — Reported as infection - unknown source
Diarrhoea (Gastrointestinal disorders) | 1
Fall (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Heart Failure (Cardiac disorders) | 1
Nervous system disorders - other (Nervous system disorders) | 1 — Neurological event and choreiform movements
Hypothyroidism (Endocrine disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=28)
Cystitis Noninfective (Renal and urinary disorders) | 6
Haematuria (Renal and urinary disorders) | 9
Hypertension (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 14
Fever (General disorders) | 3
Hypothyroidism (Endocrine disorders) | 4
Constipation (Gastrointestinal disorders) | 10
Urinary frequency (Renal and urinary disorders) | 16
Chills (General disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 9
Oedema Limbs (Skin and subcutaneous tissue disorders) | 4
Platelet Count Decreased (Blood and lymphatic system disorders) | 4
Fall (General disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 3
Nausea (Gastrointestinal disorders) | 6
Alanine Aminotransferase Increased (Gastrointestinal disorders) | 4
Urinary Tract Pain (Renal and urinary disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 3
Insomnia (General disorders) | 3
Parasthesia (Nervous system disorders) | 3
Tinnitus (Nervous system disorders) | 3
Urinary Urgency (Renal and urinary disorders) | 3
Abdominal Pain (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Renal and urinary disorders) | 2
Headache (General disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 2
Weight loss (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT02662062/Prot_SAP_000.pdf